CLINICAL TRIAL: NCT03988803
Title: A Study to Investigate the Effects of Memantine on the Pharmacokinetics of BI 425809 and Vice Versa in Healthy Male and Female Subjects (Non-randomized, Single-arm, Open-label, Three-period, One Fixed Sequence Cross-over Study)
Brief Title: A Study in Healthy Men and Women to Test Which Effects Memantine and BI 425809 Have on Each Other
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1346-0039; 2019-000468-36 (EudraCT Number)
Record Dates: First submitted 2019-06-14; First posted 2019-06-17 (Actual); Results first posted 2021-03-17 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — BI 425809; Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental)
  Interventions: Drug: BI 425809; Drug: Memantine

INTERVENTIONS:
Drug: BI 425809 — Film coated tablet
Drug: Memantine — Film coated tablet

SUMMARY:
Investigate the effect of steady state exposures of memantine on the steady-state pharmacokinetics of BI 425809 and vice versa in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation
* Male subjects, or female subjects who meet any of the following criteria from the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception that does not contain hormones, i.e. nonhormonal intrauterine device plus condom
  * Sexually abstinent
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with levels of FSH above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-randomised, single-arm, open-Label, three-period, one fixed sequence cross-over Study to investigate the effects of memantine in steady state on the pharmacokinetics of BI 425809 in steady state and vice versa in healthy male and female subjects.
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects visited specialist site to ensure that they met all implemented inclusion criteria. Subjects meeting the exclusion criteria were excluded.
Groups:
- BI 425809/Memantine/BI 425809+Memantine: Treatment period 1 (Reference 1 (R1)): Oral administration of 25 milligram (mg) BI 425809 (1 tablet of 25 mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours once daily for days 1 - 10 of period 1. Treatment period 2 (Reference 2 (R2)): Oral administration of 1 film-coated tablet of Memantine alone with 240 mL of water after an overnight fast of at least 10 hours once daily. Dose was up-titrated starting with one tablet of 5 mg for days 1-7, for days 8 -14 one tablet of 10 mg, for days 15-21 one tablet of 15 mg, for days 22 - 28 one tablet of 20 mg, and from days 29 - 35 of period 2 one tablet of 20 mg for period 2. Treatment Period 3 (Test (T)): Oral administration of 25 mg BI 425809 in combination with oral administration one tablet of 20 mg memantine with 240 mL of water after an overnight fast of at least 10 hours once daily for days 1 - 10 of period 3. Periods 1 and 2 with a washout period of at least 7 days. Period 3 followed directly after Period 2.
Period: Screening
Arm/Group | BI 425809/Memantine/BI 425809+Memantine
Started | 16
Completed | 16
Not Completed | 0
Period: Period 1
Arm/Group | BI 425809/Memantine/BI 425809+Memantine
Started | 16
Completed | 16
Not Completed | 0
Period: Period 2
Arm/Group | BI 425809/Memantine/BI 425809+Memantine
Started | 16
Treated | 15
Started Days 1 - 7: Multiple Doses of 5 mg Memantine qd | 15
Started Days 8 - 14: Multiple Doses of 10 mg Memantine qd | 14
Started Days 15 - 21: Multiple Doses of 15 mg Memantine qd | 13
Started Days 22 - 35: Multiple Doses of 20 mg Memantine qd | 13
Completed | 13
Not Completed | 3
Not completed — Prematurely discontinued from medication | 2
Not completed — Adverse Event | 1
Period: Period 3
Arm/Group | BI 425809/Memantine/BI 425809+Memantine
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were treated with at least one dose of study drug. The treated set was used for safety analyses
Arm/Group | BI 425809/Memantine/BI 425809+Memantine
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval τ (BI 425809 + Memantine : BI 425809)
Description: Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss). Comparison of BI 425809 + Memantine versus BI 425809.
  Period 1 (BI 425809):
  Measurements of steady state concentration where taken 10 minutes (min) before the next dosing of BI 425809 and 30 min, 1h, 2h, 3h, 3h 30min, 4h, 4h 30min, 5h, 6h, 7h, 8h, 10h, 12h, 24h (10 minutes (min) before the next dosing ) after first administration of BI 425809 on day 10 of Period 1.
  Treatment Period 3 (Memantine + BI 425809) Measurements of steady state concentration where taken 10 min before the next dosing of BI 425809 + Memantine and 30 min, 1h, 2h, 3h, 3h 30min, 4h, 4h 30min, 5h, 6h, 7h, 8h, 10h, 12h, 24h after first administration of BI 425809 + Memantine on day 10 of Period 3.
Time Frame: Detailed time frame is described in the measure description section.
Population: Pharmacokinetic parameter analysis set (PKS): This set included all subjects in the treated set (TS) who provided at least one pharmacokinetic (PK) endpoint that was defined as Primary and was not excluded due to protocol deviations relevant to the evaluation of PK or due to PK non-evaluability
Measure: Geometric Mean (Standard Error); unit: nanomol * hours per liter
Groups:
- BI 425809: Oral administration of 25 milligram (mg) BI 425809 (1 tablet of 25 mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours once daily for days 1 - 10 of period 1.
- Memantine + BI 425809: Oral administration of 25 milligram (mg) BI 425809 (1 tablet of 25 mg) in combination with oral administration of 1 tablet of 20 mg Memantine with 240 milliliter (mL) of water after an overnight fast of at least 10 hours for days 1 - 10 of period 3.
Arm/Group | BI 425809 | Memantine + BI 425809
Number analyzed (Participants) | 16 | 13
nanomol * hours per liter | 9029.04 (1.09) | 8559.78 (1.09)
Statistical Analysis 1: Comparison: BI 425809 vs Memantine + BI 425809; The statistical model used for the analysis of the primary endpoints was an analysis of variance (ANOVA) model on the logarithmic scale. That was, the PK endpoints were logtransformed (natural logarithm) prior to fitting the ANOVA model. The model used included effects accounting for the following sources of variation: subjects and treatment. The effect 'subjects' was considered as random, whereas the effect 'treatment' was considered as fixed; Test type: Other; ANOVA; Ratio of the geometric means (T/R1) = 94.80, 90% CI 2-sided [87.14 to 103.14], Standard Error of Mean 12.2 — Standard error of the mean is the geometric coefficient of variation

2. Primary Outcome: Maximum Measured Concentration of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval τ (BI 425809 + Memantine : BI 425809)
Description: Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss). Comparison of BI 425809 + Memantine versus BI 425809.
  Period 1 (BI 425809):
  Measurements of steady state concentration where taken 10 minutes (min) before the next dosing of BI 425809 and 30 min, 1h, 2h, 3h, 3h 30min, 4h, 4h 30min, 5h, 6h, 7h, 8h, 10h, 12h, 24h (10 minutes (min) before the next dosing ) after first administration of BI 425809 on day 10 of Period 1.
  Treatment Period 3 (Memantine + BI 425809) Measurements of steady state concentration where taken 10 min before the next dosing of BI 425809 + Memantine and 30 min, 1h, 2h, 3h, 3h 30min, 4h, 4h 30min, 5h, 6h, 7h, 8h, 10h, 12h, 24h after first administration of BI 425809 + Memantine on day 10 of Period 3.
Time Frame: Detailed time frame can be found in the measure description.
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomol per liter
Arm/Group | BI 425809 | Memantine + BI 425809
Number analyzed (Participants) | 16 | 13
nanomol per liter | 535.03 (1.07) | 531.49 (1.07)
Statistical Analysis 1: Comparison: BI 425809 vs Memantine + BI 425809; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of the geometric means (T/R1) = 99.34, 90% CI 2-sided [91.22 to 108.18], Standard Error of Mean 12.3 — Standard error fo the mean is the geometric coefficient of variation

3. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval τ (BI 425809 + Memantine : Memantine)
Description: Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss). Comparison of BI 425809 + Memantine versus BI 425809.
  Treatment Period 2 (Memantine):
  Measurements of steady state concentration where taken 10 minutes (min) before the next dosing of Memantine and 30 min, 1h, 2h, 3h, 3h 30min, 4h, 4h 30min, 5h, 6h, 7h, 8h, 10h, 12 h after administration of Memantine on day 35 of Period 2.
  Treatment Period 3 (Memantine + BI 425809) Measurements of steady state concentration where taken 10 minutes (min) before the next dosing of BI 425809 + Memantine and 30 min, 1h, 2h, 3h, 3h 30min, 4h, 4h 30min, 5h, 6h, 7h, 8h, 10h, 12h, 24h after administration of BI 425809 + Memantine on day 10 of Period 3.
Time Frame: Detailed time frame is described in the measure description section.
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomol * hours per liter
Groups:
- Memantine: Treatment period 2 (Reference 2 (R2)): Oral administration of 1 film-coated tablet of Memantine alone with 240 milliliter (mL) of water after an overnight fast of at least 10 hours once daily.
  Memantine was up-titrated starting with one tablet of 5 mg for days 1-7 of period 2, for days 8 -14 of period 2 one tablet of 10 mg Memantine daily, for days 15-21 one tablet of 15 mg Memantine daily, for days 22 - 28 of period 2 one tablet of 20 mg daily, and from days 29 - 35 of period 2 one tablet of 20 mg daily.
Arm/Group | Memantine | Memantine + BI 425809
Number analyzed (Participants) | 13 | 13
nanomol * hours per liter | 1800.36 (1.09) | 1866.76 (1.09)
Statistical Analysis 1: Comparison: Memantine vs Memantine + BI 425809; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of the geometric means (T/R2) = 103.69, 90% CI 2-sided [99.99 to 107.52], Standard Error of Mean 5.2 — Standard error fo the mean is the geometric coefficient of variation

4. Primary Outcome: Maximum Measured Concentration of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval τ (BI 425809 + Memantine : Memantine)
Description: Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss). Comparison of BI 425809 + Memantine versus BI Memantine.
  Treatment Period 2 (Memantine):
  Measurements of steady state concentration where taken 10 minutes (min) before the next dosing of Memantine and 30 min, 1h, 2h, 3h, 3h 30min, 4h, 4h 30min, 5h, 6h, 7h, 8h, 10h, 12 h after administration of Memantine on day 35 of Period 2.
  Treatment Period 3 (Memantine + BI 425809) Measurements of steady state concentration where taken 10 minutes (min) before the next dosing of BI 425809 + Memantine and 30 min, 1h, 2h, 3h, 3h 30min, 4h, 4h 30min, 5h, 6h, 7h, 8h, 10h, 12h, 24h after administration of BI 425809 + Memantine on day 10 of Period 3.
Time Frame: Detailed time frame can be found in the measure description.
Population: Pharmacokinetic parameter analysis set (PKS): This set included all subjects in the treated set (TS) who provided at least one PK endpoint that was defined as Primary and was not excluded due to protocol deviations relevant to the evaluation of PK or due to PK non-evaluability
Measure: Geometric Mean (Standard Error); unit: nanomol per liter
Arm/Group | Memantine | Memantine + BI 425809
Number analyzed (Participants) | 13 | 13
nanomol per liter | 87.06 (1.08) | 93.54 (1.08)
Statistical Analysis 1: Comparison: Memantine + BI 425809; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of the geometric means (T/R2) = 107.45, 90% CI 2-sided [102.66 to 112.45], Standard Error of Mean 6.5 — Standard error fo the mean is the geometric coefficient of variation

ADVERSE EVENTS:
Time Frame: Adverse events of BI 425809: up to 17 days. Adverse events of Memantine: up to 41 days. Adverse events of Memantine + BI 425809: up to 25 days. All-Cause Mortality was collected for up to 91 days.
Description: Treated set (TS): The treated set included all subjects who were treated with at least one dose of study drug. The treated set was used for safety analyses
Groups:
- BI 425809: Treatment period 1 (Reference 1 (R1)): Oral administration of 25 milligram (mg) BI 425809 (1 tablet of 25 mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours once daily for days 1 - 10 of period 1.
Arm/Group | BI 425809 | Memantine | Memantine + BI 425809
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 10/16 | 10/15 | 10/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 425809 (N=16) | Memantine (N=15) | Memantine + BI 425809 (N=15)
Headache (Nervous system disorders) | 5 | 4 | 2
Dizziness (Nervous system disorders) | 2 | 2 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 1
Head discomfort (Nervous system disorders) | 1 | 0 | 0
Fatigue (General disorders) | 5 | 2 | 2
Vessel puncture site reaction (General disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Change in sustained attention (Psychiatric disorders) | 0 | 0 | 1
Emotional disorder (Psychiatric disorders) | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0
Listless (Psychiatric disorders) | 1 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 1
Photophobia (Eye disorders) | 1 | 0 | 0
Eosinophil percentage increased (Investigations) | 0 | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT03988803/SAP_000.pdf
  • Study Protocol (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT03988803/Prot_001.pdf